CLINICAL TRIAL: NCT02829034
Title: A Randomized, Double-blind, Placebo Controlled, Multi-center Study to Assess the Effect of Ranolazine in Subjects With Pulmonary Hypertension and Right Ventricular Dysfunction Using Cardiovascular MRI
Brief Title: Targeting Right Ventricle in Pulmonary Hypertension Gilead
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Brigham and Women's Hospital (Other); University of Maryland (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 824808
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; right ventricular function; ranolazine
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ranolazine (Active Comparator): Ranolazine 500mg by mouth twice per day and after two weeks increase to 1000mg by mouth twice per day
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo by mouth twice per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine 500mg by mouth twice per day and after two weeks increases to 1000mg by mouth twice per day and continue for a total of 26 weeks.
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Placebo by mouth twice per day for a total of 26 weeks
  Arms: Placebo

SUMMARY:
This study is looking to see if giving ranolazine to subjects on stable pulmonary hypertension therapies but with right ventricular dysfunction (RVEF <45%) will improve their health by improving right ventricular (RV) function.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pulmonary hypertension based on one of the following criteria:

  * Idiopathic pulmonary arterial hypertension
  * Familial pulmonary arterial hypertension
  * Pulmonary hypertension associated with connective tissue disease
  * Chronic thromboembolic pulmonary hypertension-nonsurgical/distal vessel disease or patients who are reluctant to go to surgery within a 6-month period and are willing to participate
  * Simple congenital such as repaired atrial septal defect or ventricular septal defect or unrepaired small atrial septal defect or ventricular septal defect with persistent and out of proportion pulmonary arterial hypertension
  * Group 3 patients who have a component of pulmonary arterial hypertension *Pulmonary hypertension caused by conditions affect the veins and small vessels of the lungs
  * Sickle cell disease
  * Group 5 pulmonary hypertension such as polycythemia vera
  * Essential thrombocythemia
  * Sarcoidosis
  * Vasculitis
  * Metabolic disorder
* World Health Organization functional class II, III, or IV
* Mean pulmonary artery pressure >25 mmHg at rest
* Pulmonary capillary wedge pressure or left ventricular end diastolic pressure < 15 mmHg
* Pulmonary vascular resistance > 3 mmHg/L/min
* Right ventricle ejection fraction < 45%
* 6-minute walk test distance > 50 meters

Exclusion Criteria:

* Previous treatment with or prior sensitivity to ranolazine
* Any family history of corrected QT interval prolongation, congenital long QT syndrome, or receiving drugs that prolong the corrected QT interval
* Parenchymal lung disease showing total lung capacity < 50% of predicted OR forced expiratory volume at one second/forced vital capacity < 50%
* Portal hypertension associated with chronic liver disease
* Left sided heart disease including any of the following: moderate or greater aortic or mitral valve disease, Any left ventricle cardiomyopathy, Left ventricular systolic dysfunction defined as an ejection fraction < 50%, Symptomatic coronary artery disease
* Uncontrolled systemic hypertension
* Implantable cardioverter-defibrillator, Pacemaker, hazardous metallic implants or any other contraindication to MRI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Han, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han Y, Forfia PR, Vaidya A, Mazurek JA, Park MH, Ramani G, Chan SY, Waxman AB. Rationale and design of the ranolazine PH-RV study: a multicentred randomised and placebo-controlled study of ranolazine to improve RV function in patients with non-group 2 pulmonary hypertension. Open Heart. 2018 Feb 23;5(1):e000736. doi: 10.1136/openhrt-2017-000736. eCollection 2018. PMID 29531764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 14 | 8
Completed | 9 | 6
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 14 | 8 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 20
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (16.9) | 53.6 (14.1) | 54.8 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline Right Ventricular Ejection Fraction (the Unit is Percentage)
Description: Change in right ventricle ejection fraction as assessed by MRI
Time Frame: 26 weeks
Population: participants who completed follow up study at 6 months.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 9 | 6
percentage | 7.56 (1.72) | -3.99 (2.23)

2. Secondary Outcome: Percent Change in 6min-walk-test Distance
Description: 6-minute walk test
Time Frame: 6 months
Population: complete and recorded data
Measure: Least Squares Mean (Standard Error); unit: percentage of distance walked
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 8 | 5
percentage of distance walked | -0.09 (0.095) | -0.06 (0.125)

3. Secondary Outcome: Change in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP measured at 6-months compared to baseline
Time Frame: 6 months
Population: completers
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 9 | 6
pg/mL | -119.72 (276.42) | -287.75 (353.81)

ADVERSE EVENTS:
Time Frame: 7 months including 6 months of drug treatment and 1 month post treatment
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/8
Serious Adverse Events (participants affected / at risk) | 3/14 | 2/8
Other Adverse Events (participants affected / at risk) | 11/14 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=14) | Placebo (N=8)
heart failure (Cardiac disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=14) | Placebo (N=8)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
dark urine (Renal and urinary disorders) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
leg weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
restless sleep (Nervous system disorders) | 1 (1) | 0 (0)
dryness on CPAP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TENOSYNOVITIS, (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
fatique (General disorders) | 1 (1) | 0 (0)
bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT02829034/Prot_SAP_000.pdf